CLINICAL TRIAL: NCT06025929
Title: Effectiveness of Maitland Mobilization Versus Mulligan Mobilization Techniques With Common Use of Interferential Therapy in Patients With Knee Joint Osteoarthritis
Brief Title: Effect of Different Mobilization Techniques With Common Use of Interferential Therapy in Patients With Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Burdwan Institute of Medical and Life Sciences (BIMLS) (Unknown)
Responsible Party: Principal Investigator, AMIR IQBAL, Prinicipal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIMLS/67/2017
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis
Keywords: Maitland mobilization; Mulligan mobilization; Knee pain; Interferential therapy; WOMAC; Functional limitation
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland Group (Experimental): Maitland Group received Maitland's mobilization techninque in addition to an intereferential therapy.
  Interventions: Other: Maitland's mobilization technique; Other: Interferential Therapy (IFT)
- Mulligan Group (Active Comparator): Mulligan Group received Mulligan's mobilization techninque in addition to an intereferential therapy.
  Interventions: Other: Mulligan's mobilization techniques; Other: Interferential Therapy (IFT)

INTERVENTIONS:
Other: Maitland's mobilization technique — Maitland's mobilization technique was performed on the patients with its all components, such as 1. Distraction 2. Anteroposterior glides 3. Posteroanterior glides 4. Medial glides and 5. Lateral glides.
  Arms: Maitland Group
Other: Mulligan's mobilization techniques — Mulligan's mobilization technique was performed on the patients with its all components using a therapeutic belt, such as 1. Medial mobilization with movement (MWM) for Knee flexion 2. Medial mobilization with movement (MWM) for Knee extension 3. Lateral mobilization with movement (MWM) for Knee flexion 4. Lateral mobilization with movement (MWM) for Knee extension.
  Arms: Mulligan Group
Other: Interferential Therapy (IFT) — Interferential Therapy was performed on the patients with the following parameters: career frequency 4000Hz; waveform: rectangular; sweep time: 1 second rise and fall and 5 second stay; Treatment duration: 10 minutes; sweep frequency: 10 to 130 Hz. The current intensity was adjusted until the subject reported feeling a strong tingling sensation without causing muscle contraction. A aquatic gel was applied before straping the electopads over treatment area for smooth electrical conduction.

SUMMARY:
This study aimed to determine the effects of different manual mobilization techniques on pain, muscle strength, and functional limitations in individuals with knee osteoarthritis (Knee OA). A double-blinded pretest-posttest experimental study. This research employed a two-arm parallel group randomized comparative design. A total of thirty participants diagnosed with knee osteoarthritis were randomly assigned and equally divided into groups 1 and 2, each containing 15 participants. Both Group 1 and Group 2 underwent Maitland and Mulligan mobilization techniques, alongside a common Interferential therapy (IFT) regimen, over the course of three sessions per week for a duration of four weeks. The assessment of pain and functional disability outcomes was conducted through the application of The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores at the baseline and four weeks following the intervention. To determine the effects of the intervention within and between the groups, the outcome scores were subjected to analysis using both dependent and independent t-tests.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a prevalent disorder with significant global health implications, its prevalence varying across populations due to intricate factors. Recent investigations highlight an age-related increase in knee OA prevalence, particularly impacting those aged 60 and above, with projections indicating heightened impact due to aging demographics. Recent pathogenesis studies illuminate the intricate molecular and cellular processes underlying knee osteoarthritis (OA), encompassing cartilage degradation, subchondral bone changes, and inflammation.Recent advancements have expanded knee osteoarthritis (OA) management, including medical, surgical, and physiotherapy interventions. Pharmacological treatments such as analgesics, non-steroidal anti-inflammatory drugs (NSAIDs), and disease-modifying osteoarthritis drugs (DMOADs) remain fundamental for pain alleviation and inflammation reduction. Intra-articular therapies like corticosteroid injections and hyaluronic acid supplements offer localized relief and potential disease-modifying effects.Surgical interventions like total knee arthroplasty (TKA) provide pain relief and improved function for end-stage OA. Minimally invasive techniques like partial knee replacements and patient-specific implants aim to preserve joint function and enhance outcomes. Physiotherapy and rehabilitation are crucial, in improving stability, muscle strength, and mobility. Studies highlight tailored exercises, neuromuscular training, and proprioceptive exercises in managing OA symptoms. The integration of these approaches underscores comprehensive knee OA management, addressing pain, function, and quality of life. The outcomes of this study could offer evidence-based recommendations for clinicians, aiding them in selecting the most appropriate manual therapy approach to alleviate pain, enhance joint mobility, and improve functional capacity in knee OA patients. Ultimately, this research seeks to contribute to the optimization of knee OA management strategies, improving the well-being of those affected.

ELIGIBILITY:
Inclusion Criteria:

* Sub-acute or chronic osteoarthritis of knee.
* Age between 45-65 years.
* Gender Male and female.
* Subjects willing to participate in the study

Exclusion Criteria:

* Presence of R.A, polyarthritis or systemic inflammatory arthropathies.
* History of total knee arthroplasty or major knee trauma injury.
* Fracture of lower limb within the past 6 months.
* Hip or ankle instability, excessive weakness, surgery or major trauma injury.
* Intra-articular steroid injection in knee joint within 3 months.
* Cognitive problems.
* Patient with severe cardiac or pulmonary disorders.
* Peripheral vascular disease.
* Tumour/malignancies/infections.
* Metallic implants in the lower limbs.
* Any severe deformity around the knee joint.
* Kellgren and Lawrence (KL) system47: up to grade 0-III.
* History of neurological and psychological disorders.
* High risk health status- e.g.- uncontrolled hypertension, diabetes, heart disease, angina type pain, nocturnal dyspnoea, shortness of breathing, tachycardia etc.
* Contraindications of IFT and mobilization.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Functional limitations | 4 weeks
  Functional limitations was assessed using the Western Ontario and McMaster Universities (WOMAC) index. It includes five questions about pain, two about stiffness, and 17 on degree of disability of activities of daily living. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT, Study Chair — King Saud University
Locations (1):
- Department of Rehabilitation Sciences, College of applied Medical Science, King Saud University, Riyadh, Saudi Arabia